CLINICAL TRIAL: NCT07087379
Title: Perioperative Intensive Statin Therapy for Neuroprotection in Transcatheter Aortic Valve Replacement
Brief Title: Perioperative Intensive Statin Therapy for Neuroprotection in TAVR（PISTNT）
Acronym: PISTNT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pan Xiangbin (Other)
Responsible Party: Sponsor-Investigator, Pan Xiangbin, Vice President of Fuwai Hospital, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025-055-01; 2025YFKT-ZL-09 (Other Grant/Funding Number: Fuwai Yunnan Hospital, Chinese Academy of Medical Sciences)
Record Dates: First submitted 2025-07-17; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Aortic Stenosis; Cerebral Ischaemic Injury
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Statin Group (Experimental)
  Interventions: Drug: Intensive statin treatment
- Controll Group (Placebo Comparator)
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: Intensive statin treatment — Intensive statin group:
  Atorvastatin 80mg, orally administered 12 hours before surgery Atorvastatin 80mg, orally administered 2 hours before surgery
  Arms: Intensive Statin Group
Drug: Placebo Control — Placebo, tablets, oral administration 12 hours before surgery Placebo, tablet, oral administration 2 hours before surgery
  Arms: Controll Group

SUMMARY:
Transcatheter aortic valve replacement (TAVR) has become the most anticipated treatment method in the cardiovascular field in recent years, experiencing rapid development. However, neurological complications related to the surgery, such as ischemic injury, stroke, transient ischemic attack, and postoperative delirium, remain the main causes of increased postoperative mortality. Currently, there are limited measures for neuroprotection during the perioperative period of TAVR, and controversy continues over the effectiveness of intraoperative cerebral device placement. Consequently, strategies for neuroprotection during TAVR require active exploration. Previous studies have shown that statins have pleiotropic effects. In addition to inhibiting cholesterol synthesis, it also exhibits anti-inflammatory, antioxidant, stress-reducing, and platelet aggregation-inhibiting properties, as well as potential neuroprotective effects. The efficacy and safety of intensive statin therapy during the perioperative period of percutaneous coronary intervention have been extensively examined, and its role in improving long-term prognosis has been recognised. Since coronary heart disease and aortic valve stenosis share similar pathophysiological mechanisms, the use of statins in valve replacement surgery has also demonstrated positive effects. Research indicates that preoperative high-intensity statin therapy can reduce the incidence of stroke or transient ischemic attack following valve replacement surgery. Additionally, evidence suggests that preoperative statin use can decrease the occurrence of postoperative delirium. However, no evidence exists on whether perioperative intensive statin therapy during TAVR can reduce cerebral ischaemic injury and provide neuroprotection. This study aims to conduct a prospective, randomised, double-blind, multicentre clinical trial to evaluate the neuroprotective effects of statin-enhanced therapy during the perioperative period of TAVR and to investigate whether it can reduce cerebral ischaemic injury after TAVR.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥65-80 years with symptomatic severe aortic stenosis at the time of screening for enrollment;
* It is planned to undergo transcatheter aortic valve replacement at a scheduled time;
* Informed consent from the patient or the guardian;
* American Society of Anesthesiologists (ASA) classification I-III;
* Possess comprehensive reading, listening, and speaking abilities, and be able to cooperate in completing neuropsychological tests

Exclusion Criteria:

* Impaired preoperative cognitive function, with a Montreal Cognitive Assessment score of ≤20;
* Previous history of disabling stroke (modified Rankin Scale score ≥3) or carotid stenosis exceeding 70%, or severe stenosis of the subclavian artery or brachiocephalic trunk;
* Preoperative baseline MRI indicated acute or subacute ischemic brain injury;
* Have taken statins within the past month;
* Renal failure (glomerular filtration rate (GFR) <30 mL/min/1.73 m2);
* Allergic to atorvastatin;
* Contraindications to atorvastatin (active liver disease with unexplained persistent elevation of liver enzymes/history of muscle disease);
* Patients with permanent pacemaker implantation or those who cannot undergo MRI due to claustrophobia;
* Severe systemic disease with an expected life expectancy of less than 90 days;
* There are any other medical or non-medical reasons, such as inability to comply with research procedures or follow-up, or plans to relocate during the study period, that the researcher deems unsuitable for the subject to participate in the study

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
The number of new ischemic lesions on brain DW-MRI on the third day after TAVR | Day 3
  Compared to baseline DW-MRI, the number of newly discovered cerebral ischemic lesions in the subjects on the third day after randomization and surgery, as assessed by cranial DW-MRI scans.